CLINICAL TRIAL: NCT02726282
Title: Impact of Papillary Microcarcinoma Terminology on Patients Treatment Preferences
Brief Title: Impact of Papillary Microcarcinoma Terminology on Patients Treatment Preferences: a Cross Sectional Survey
Status: Withdrawn | Type: Observational
Why Stopped: funding not available
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juan P. Brito Campana, MBBS, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 15-008166
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To explore how a clinical sample of patients with thyroid nodules (men and women) with no history of thyroid cancer would make decisions about treatments based on different terminology used to describe papillary thyroid cancer (with and without the cancer term).

ELIGIBILITY:
Inclusion Criteria:

* able to complete a survey

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of thyroid nodules
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Treatment choice | one year

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Brito, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States